CLINICAL TRIAL: NCT03516019
Title: Messaging Intervention Trial in the Electronic Framingham Heart Study (eFHS)
Brief Title: eFHS Messaging Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: H-36586; 74624 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Diseases
Keywords: mHealth; digital BP monitoring; patient provider communication; smart watch; user engagement; population health data
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The research design includes a cohort eFHS Study and an embedded randomized factorial trial on a subset of the cohort.
Who Masked: Investigator
Masking Description: eFHS researchers, statistician, research assistant, and clinic staff are masked to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Weekday am personalized notices (Experimental): Participants in this arm receive personalized weekday am notices on Wednesday at 7am.
  Interventions: Other: personalized notices; Other: am notices; Other: weekday notices
- Weekday pm personalized notices (Experimental): Participants in this arm receive a personalized weekday pm notices on Wednesday at 7pm.
  Interventions: Other: personalized notices; Other: pm notices; Other: weekday notices
- Weekend am personalized notices (Experimental): Participants in this arm receive a personalized weekend am notices on Saturday at 7am.
  Interventions: Other: personalized notices; Other: am notices; Other: weekend notices
- Weekend pm personalized notices (Experimental): Participants in this arm receive personalized pm notices on Saturday at 7pm.
  Interventions: Other: personalized notices; Other: pm notices; Other: weekend notices
- Weekday am standard notices (Experimental): Participants in this arm receive standard weekday notices on Wednesday at 7am.
  Interventions: Other: standard notices; Other: am notices; Other: weekday notices
- Weekday pm standard notices (Experimental): Participants in this arm receive standard weekday notices on Wednesday at 7pm
  Interventions: Other: standard notices; Other: pm notices; Other: weekday notices
- Weekend am standard notices (Experimental): Participants in this arm receive standard weekend notices on Saturday at 7am
  Interventions: Other: standard notices; Other: am notices; Other: weekend notices
- Weekend pm standard notices (Experimental): Participants in this arm receive standard weekend notices on Saturday at 7pm
  Interventions: Other: standard notices; Other: pm notices; Other: weekend notices

INTERVENTIONS:
Other: personalized notices — The personalized notices take into account if data were received over the previous week, and accordingly encourages the participant to use the device and send her data, or encourages the participant to continue using the device and sending data. A library of personalized notices with alternative motivational content was developed. Each time a notification is sent, it will be drawn at random from the library.
  Arms: Weekday am personalized notices; Weekday pm personalized notices; Weekend am personalized notices; Weekend pm personalized notices
Other: standard notices — The standard notices which are neutral and invite participants to wear the watch daily and to measure their blood pressure weekly.
  Arms: Weekday am standard notices; Weekday pm standard notices; Weekend am standard notices; Weekend pm standard notices
Other: am notices — notifications sent at 7 am.
  Arms: Weekday am personalized notices; Weekday am standard notices; Weekend am personalized notices; Weekend am standard notices
Other: pm notices — notifications sent at 7 pm.
  Arms: Weekday pm personalized notices; Weekday pm standard notices; Weekend pm personalized notices; Weekend pm standard notices
Other: weekday notices — notifications sent on Wednesday
  Arms: Weekday am personalized notices; Weekday am standard notices; Weekday pm personalized notices; Weekday pm standard notices
Other: weekend notices — notifications sent on Saturday
  Arms: Weekend am personalized notices; Weekend am standard notices; Weekend pm personalized notices; Weekend pm standard notices

SUMMARY:
In this research the investigators will develop and test an innovative scalable mobile health and digital cardiovascular monitoring system within a longitudinal deeply characterized cohort with three components: 1) smartphone application (app) designed to promote adherence, integrate digital and mHealth information, and facilitate communication with participants and researchers; 2) smartwatch activity monitoring using the Apple iWatch; and 3) home blood pressure (BP) monitoring using the Withings blood pressure device.

The objective of the messaging trial is to test the effect of messaging strategies on improving participants' long-term use of and engagement with our selected mobile health technologies and on increasing response rate of survey data collection.

DETAILED DESCRIPTION:
The research design includes a cohort eFHS Study and an embedded randomized factorial trial on a subset of the cohort.

For the primary e-cohort, the investigators will build a custom mobile app for use within the Framingham Heart Study (FHS) to digitally collect data, compare it against research clinic-collected data, quantify risk factor burden, and perform CVD risk prediction. The app development will focus on 1) CVD risk factor data that would benefit from more frequent ascertainment than the every four to eight year FHS examination cycles; 2) circumstances where in vivo assessment may be superior to clinic-based assessment; 3) key endpoints of the FHS that are considered FHS landmarks. In addition to the eFHS App, participants will be offered wireless devices (Withings BP) to measure blood pressure and an Apple Watch to measure heart rate and steps per day.

For the messaging trial, the investigators will conduct a randomized factorial trial phase to test the effect of messaging strategies. Participants will be sent a weekly notification through the eFHS app. Participants will be randomly allocated to one of 8 groups defined according to the following: using personalized reminder messaging vs. standard neutral messaging; notification sent on a weekday vs. weekend; notification sent in the morning vs. the evening. The three main comparisons will be simultaneously evaluated according to a 2x2x2 factorial design.

ELIGIBILITY:
Inclusion Criteria for the eFHS study:

* Participants of the FHS Third Generation, Omni Group 2, and New Offspring Spouse Cohorts attending the in-person examination 3 with access to a smartphone or home internet access and English speaking/reading.

Specifically for the RCT substudy (re: engagement with select mobile health technologies):

* English-speaking individual
* Owns an iPhone with compatible iOS (version 9 or higher);
* Residence in the United States
* Provision of permissions for notifications and data sharing with the Research Center
* Provision of signed and dated informed consent

Exclusion Criteria:

* Participants who do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2018-05-19 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2019-03-23 (Actual)

PRIMARY OUTCOMES:
Adherence at 3 months to the weekly BP recording | 3 months
  proportion of participants who submit their weekly blood pressure measurement at 3 months
Adherence at 3 months to the weekly HR recording | 3 months
  proportion of participants who submit their weekly heart rate measurement at 3 months

SECONDARY OUTCOMES:
Adherence at one month to the weekly BP recording | 1 month
  proportion of participants who submit their weekly blood pressure measurement at 1 month
Adherence at one month to the weekly HR recording | 1 month
  proportion of participants who submit their weekly heart rate measurement at 1 month

OTHER OUTCOMES:
Adherence to survey response | 3 months
  proportion of participants who complete the eFHS survey at 3 months
Adherence at 6 months to the weekly BP recording | 6 months
  Comparison between the groups receiving personalized notices to the groups receiving standard notices
Adherence at 6 months to the weekly HR recording | 6 months
  Comparison between the groups receiving personalized notices to the groups receiving standard notices
Adherence at 6 months to survey response | 6 months
  Comparison between the groups receiving personalized notices to the groups receiving standard notices

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Murabito, MD ScM, Principal Investigator — Framingham Heart Study
Locations (1):
- Framingham Heart Study, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trinquart L, Liu C, McManus DD, Nowak C, Lin H, Spartano NL, Borrelli B, Benjamin EJ, Murabito JM. Increasing Engagement in the Electronic Framingham Heart Study: Factorial Randomized Controlled Trial. J Med Internet Res. 2023 Jan 20;25:e40784. doi: 10.2196/40784. PMID 36662544